CLINICAL TRIAL: NCT01197469
Title: Do Phosphodiesterase 5A Inhibitors Improve Exercise Capacity in Patients With Chronic Obstructive Pulmonary Disease and Pulmonary Hypertension?
Brief Title: Do Phosphodiesterase 5A Inhibitors Improve Exercise Capacity in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Pulmonary Hypertension?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government); NHS Tayside (Other Government); NHS Fife (Other Government)
Responsible Party: Principal Investigator, A. D. Struthers, Chief Investigator, University of Dundee
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2008CV17
Record Dates: First submitted 2010-09-01; First posted 2010-09-09 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Hypertension
Keywords: Secondary Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Tadalafil (Active Comparator)
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — Tadalafil 10mg once daily for 3 months
  Arms: Tadalafil
Drug: Placebo
  Arms: Placebo

SUMMARY:
The investigators hypothesise that phosphodiesterase 5A inhibitors will improve exercise capacity in those with Chronic Obstructive Pulmonary Disease and secondary pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* Forced expiratory volume in 1 second (FEV1) <80% (FEV1/FVC <0.70)
* Right ventricular systolic pressure (RVSP) > 30 mmHg or Pulmonary Acceleration time <120 ms

Exclusion Criteria:

* Pulmonary stenosis or echo left ventricular outflow tract obstruction
* Left ventricular ejection fraction < 45%
* Patients taking nitrates, nicorandil or doxazosin.
* Drug contraindications:

  * Systolic Blood Pressure <90 mmHg
  * recent stroke
  * unstable angina
  * past history of non arteritic anterior ischaemic optic neuropathy

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
6 minute walking distance | 3 months
  The investigators will perform a baseline 6 minute walking distance (0 months) and repeat the measure at 2 months and finally at 3 months

SECONDARY OUTCOMES:
Quality of Life | 3 months
  The investigators will measure baseline quality of life (0 months) using St George's Respiratory Questionnaire, SF-36v2, Minnesota Heart Failure Questionnaire. These questionnaires will be repeated at 2 and 3 months (final measurement).
B- Natriuretic Peptide (BNP) | 3 months
  Will be measured at 0, 2 and 3 months
Diffusion lung capacity for carbon monoxide (DLCO) | 3 months
  Will be measured at 0 and 3 months
Echocardiographic measurements | 3 months
  Will be measured at 0 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan Struthers, MBChB, Principal Investigator — University of Dundee
Locations (1):
- University of Dundee, Dundee, Tayside, United Kingdom

REFERENCES:
- [Derived] Goudie AR, Lipworth BJ, Hopkinson PJ, Wei L, Struthers AD. Tadalafil in patients with chronic obstructive pulmonary disease: a randomised, double-blind, parallel-group, placebo-controlled trial. Lancet Respir Med. 2014 Apr;2(4):293-300. doi: 10.1016/S2213-2600(14)70013-X. Epub 2014 Mar 5. PMID 24717626